CLINICAL TRIAL: NCT04874818
Title: [89Zr]Df-IAB22M2C Anti-CD8 Minibody PET/CT Imaging to Assess the in Vivo Distribution of CD8+ T-cells in COVID-19 Patients
Brief Title: CD8+ T-cell PET/CT Imaging in COVID-19 Patients
Acronym: Tangelo
Status: Terminated | Type: Observational
Why Stopped: COVID-19 pandemic resided
Sponsor: Radboud University Medical Center (Other)
Collaborators: ImaginAb, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NL76248.091.20; 2020-005984-29 (EudraCT Number)
Record Dates: First submitted 2021-04-28; First posted 2021-05-06 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-06

CONDITIONS: Lymphopenia Due to COVID-19; T-cell; PET Imaging
Keywords: COVID-19; lymphopenia; T-cells; PET imaging
MeSH Terms: conditions — COVID-19; Lymphopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- lymphopenia: lymphocyte counts (<1.0 x10e9/L)
  Interventions: Diagnostic Test: [89Zr]Df-IAB22M2C PET/CT scan
- normal lymphocyte numbers: lymphocyte counts ((1.0 - 3.5 x10e9/L))
  Interventions: Diagnostic Test: [89Zr]Df-IAB22M2C PET/CT scan

INTERVENTIONS:
Diagnostic Test: [89Zr]Df-IAB22M2C PET/CT scan — PET imaging procedure

SUMMARY:
A subset of patients diagnosed with severe acute respiratory syndrome (SARS)-CoV2 infection present with lymphopenia. The degree of lymphopenia, and in particular reduced cluster of differentiation (CD)8+ T-cell numbers, is correlated with clinical deterioration and intensive care unit (ICU) admission. The underlying reasons for lymphopenia in coronavirus disease (COVID)-19 is currently unclear, We aim to assess differences in the in vivo distribution of CD8+ T-cells in patients with proven SARS-CoV2 presenting with lymphopenia or with normal lymphocyte counts, using Zirconium-89 ([89Zr])Df-IAB22M2C positron emission tomography (PET) imaging.

DETAILED DESCRIPTION:
Rationale: A subset of patients diagnosed with SARS-CoV2 infection present with lymphopenia. The degree of lymphopenia, and in particular reduced CD8+ T-cell numbers, is strongly correlated with clinical deterioration and ICU admission .

The underlying reasons for lymphopenia in COVID-19 is currently unclear, but several hypotheses have been put forward; 1) sequestration of CD8+ T-cells in peripheral tissues (e.g. lung) either during the effector phase of their lifespan or passively by local chemotactic signals, 2) accelerated maturation and apoptosis either induced by storm of inflammatory cytokines or direct infection or 3) resulting from decreased lymphopoiesis induced by reduced levels of stem cell factor. The lack of data on in vivo distribution of CD8+ T-cells hampers a more thorough understanding of this critical prognostic factor.

Aim: We aim to assess differences in the in vivo distribution of CD8+ T-cells in patients with proven SARS-CoV2 presenting with lymphopenia or with normal lymphocyte counts, using [89Zr]Df-IAB22M2C PET/CT imaging.

Study design: This is a prospective, observational non-randomized pilot study in 20 patients with microbiologically proven SARS-CoV2 infection. All patients will undergo a whole body [89Zr]Df-IAB22M2C PET/CT scan.

Study population: Twenty patients ≥50 years of age with proven COVID-19, who are admitted to the ward will be included, patients will be stratified according to lymphocyte counts on admission to ensure an even distribution: presenting with lymphopenia (<1.0 x10e9/L) (n=10) and with lymphocyte numbers within normal range (1.0 - 3.5 x10e9/L) (n=10).

Study procedure: All patients will undergo a [89Zr]Df-IAB22M2C PET/CT scan 21-27 hours post intravenous injection of 1.5mg protein dose labelled with 37 megabecquerel (MBq) (1 mCi) 89Zr; and one additional blood sample at the day of scanning.

Primary study objective: The primary objective of this study is to assess differences in the in vivo distribution of CD8+ T-cells in patients with proven SARS-CoV-2 presenting with lymphopenia or with normal lymphocyte counts, using [89Zr]Df-IAB22M2C PET/CT imaging.

Secondary study objectives:

1. To assess the spatial correlation between [89Zr]Df-IAB22M2C uptake and abnormal findings on routine contrast-enhanced CT scan of the chest
2. To assess the correlation between in vivo biodistribution of [89Zr]Df-IAB22M2C and concurrent flowcytometric phenotypic and quantitative assessment of lymphocyte populations
3. To explore the correlation between in vivo biodistribution of [89Zr]Df-IAB22M2C and clinical course of disease

ELIGIBILITY:
Inclusion Criteria:

* a microbiologically proven SARS-CoV2 infection
* More than 50 years of age;
* Ability to provide written informed consent.

Exclusion Criteria:

* Contra-indication for PET: Pregnancy, Breast-feeding, Severe claustrophobia.
* Contra-indication for administration of iodine-containing contrast agents
* Other serious illness, e.g. history of malignancies or auto-immune disorders
* Known pre-existing lymphopenia from an unrelated other medical condition
* Estimated creatinine clearance ≤ 30 mL/min according to the Cockcroft-Gault formula (or local institutional standard method) OR oligo-uric patients (<400 mL/24hr)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population for this pilot study exists of 20 evaluable patients with a proven SARS-CoV2 infection admitted to the Infectious Diseases ward. Patients presenting in the Radboud University Medical Center will be considered for recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to quantify uptake of [89Zr]Df-IAB22M2C, as a surrogate for the presence of CD8+ T-cells, in major organ systems of patients with proven SARS-CoV-2 presenting with lymphopenia or with normal lymphocyte counts. | 18 months
  The main study parameter is the SUVmean uptake of [89Zr]Df-IAB22M2C in major organs systems, e.g. lungs, spleen, bone marrow, liver and bloodpool

SECONDARY OUTCOMES:
Based on imaging | 18 months
  1) Spatial correlation of SUVmean per lung segment with CORADS score per lung segment
Based on laboratory parameters | 18 months
  2) In vivo biodistribution of [89Zr]Df-IAB22M2C will be correlated to laboratory test 3) In vivo biodistribution of [89Zr]Df-IAB22M2C will be correlated with lymphocyte counts (x10e9/L)
Based on clinical characteristics | 18 months
  4) In vivo biodistribution of [89Zr]Df-IAB22M2C will be correlated with duration of hospital stay (days)

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud university medical center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No